CLINICAL TRIAL: NCT05778149
Title: Safety and Efficacy of Aumolertinib Combined With Anlotinib as 1st Line Treatment in Advanced Lung Cancer EGFR Mutation With TP53 Co-Mutation
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA-53
Record Dates: First submitted 2023-03-08; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Aumolertinib; Anlotinib; TP53; NSCLC; EGFR Activating Mutation
MeSH Terms: interventions — aumolertinib; anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): single arm,Treatment plan: Aumolertinib 110mg p.o QD; Anlotinib 12mg, oral for 2 weeks, three weeks a cycle, until disease progression.
  Interventions: Drug: Aumolertinib,Anlotinib

INTERVENTIONS:
Drug: Aumolertinib,Anlotinib — Aumolertinib 110mg p.o QD; Anlotinib 12mg, oral for 2 weeks, three weeks a cycle, until disease progression.

SUMMARY:
The goal of this open, single-arm, exploratory phase II clinical study is to exploratory safety and efficacy in 1st line treatment in advanced lung cancer EGFR mutation with TP53 co-mutation. 47 patients are scheduled to be enrolled. Treatment regimen is aumolertinib 110mg p.o QD and Anlotinib 12mg oral for 2 weeks, three weeks a cycle, until disease progression or intolerable adverse reactions or death.

DETAILED DESCRIPTION:
The primary objective of this study was to explore the median PFS of aumolertinib Combined With anlotinib as first-line treatment in advanced lung cancer EGFR mutation with TP53 co-mutation.The secondary objective of this study was to evaluate the ORR, DCR, DOR, OS and safety of aumolertinib Combined With anlotinib as first-line treatment in advanced lung cancer EGFR mutation with TP53 co-mutation. In addition, we also try to explore predictive or prognostic biomarkers (tissue and/or plasma) related to disease treatment response or drug resistance. Analyze the potential biomarkers in the biopsy tissue samples and blood samples after the disease progresses, and explore the possible mechanism of treating drug resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Locally advanced or metastatic NSCLC EGFR sensitive mutations (19del and L858R) and TP53 co-mutation;
2. Age 18-85 years, male or female;
3. Have not received systematic treatment; If the subject has received adjuvant therapy after completing radical treatment for early gastric cancer and the subject has relapsed disease, ensure that the end of adjuvant therapy is more than 6 months from the first dose of the study and that various toxicities due to the adjuvant therapy have recovered;
4. ECOG 0-1, The expected survival is more than 6 months;
5. At least one assessable lesion (RECIST 1.1 );
6. If the main organs function normally, they meet the following standards:

   1. Absolute value of neutrophils (ANC) ≥ 1.5 × 10 ^ 9 /L;
   2. platelet count ≥ 100 × 10 ^ 9 /L
   3. hemoglobin ≥ 90g /L;
   4. white blood cell ≥ 3.0 × 10^9\/L；
   5. Liver function: total bilirubin<1.5 times the upper limit of normal value, aspartate aminotransferase (AST /SGOT), alanine aminotransferase (ALT /SGPT) and alkaline phosphatase (ALP) ≤ 2.5 times the upper limit of normal value; In case of liver metastasis, AST and ALT ≤ 5.0 times the upper limit of normal value; In case of liver metastasis and/or bone metastasis, ALP ≤ 5.0 times the upper limit of normal value.
   6. Renal function: serum creatinine (Scr) ≤ 1.5 times the upper limit of normal value; Urine routine test: urine protein<2 (+); If the urine protein at baseline is ≥ 2 (+), the 24-hour urine protein quantity must be ≤ 1.0g;
   7. Coagulation function: international normalized ratio (INR) ≤ 1.5, and activated partial thromboplastin time (APTT) ≤ 1.5 times the upper limit of normal value;

Exclusion Criteria:

1. Squamous cell carcinoma (including adenosquamous carcinoma and undifferentiated carcinoma); Small cell lung cancer (including small cell and non-small cell mixed lung cancer); Patients who have received systemic therapy in the past (allow to receive adjuvant or neoadjuvant therapy in the past);
2. Patients with symptomatic brain metastasis at the beginning of treatment (patients with brain metastasis who have received treatment in the past are eligible if asymptomatic brain metastasis lasts for at least 4 weeks when receiving stable dose of drug treatment);
3. . Patients who participated in the intervention tumor clinical trial during the first-line treatment or within the last 30 days before the first-line treatment;
4. History of tracheoesophageal fistula, gastrointestinal perforation or gastrointestinal fistula and intra-abdominal abscess within 6 months before treatment;
5. Suffer from serious cardio-cerebrovascular disease;
6. Subjects who received chest radiotherapy in the lung field within the first 4 weeks, or who have not recovered from radiotherapy-related toxicity. Subjects who received radiotherapy or did not recover from radiotherapy-related toxicity within 2 weeks before randomization for all other anatomical sites;
7. Major surgical treatment was performed within 4 weeks before treatment or planned during the trial period (the researcher judged that there was bleeding risk or wound healing complications);
8. . Have bleeding tendency, high bleeding risk or coagulation dysfunction, including thrombotic disease within 6 months before randomization and/or hemoptysis history within 3 months before randomization (single cough bleeding ≥ 2.5mL)
9. Subjects with high suspicion of idiopathic pulmonary fibrosis, organic pneumonia, drug-related pneumonia, idiopathic pneumonia or active pneumonia on chest CT scan during screening period;
10. Imaging examination showed that there was evidence of tumor invasion into large vessels, and the tumor had completely approached, surrounded or invaded the lumen of large vessels (such as pulmonary artery or superior vena cava);
11. Subjects with hypertension (systolic blood pressure>160mmHg or diastolic blood pressure>100mmHg) that are still poorly controlled after treatment with two or more antihypertensive drugs in the screening period, and who have a history of hypertensive crisis or hypertensive brain disease in the past;
12. Those with unhealed wounds, active digestive ulcer, fractures (excluding old healed fractures);
13. Known or suspected to be allergic to aumolertinib and Anlotinib and/or other components of their preparations;
14. Pregnant or lactating women;
15. Women or male subjects of childbearing age who are unwilling to take effective contraceptive measures during the study period or within 6 months after the last administration of the study drug
16. In addition to the above conditions, the researcher believes that there are other conditions that are not suitable for selection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2023-03-31 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
PFS (Progression-Free-Survival) | 24months
  The time from randomization to tumor progression or death.The efficacy of this study was determined according to Recist version 1.1 criteria.

SECONDARY OUTCOMES:
ORR（Objective Response Rate） | 24months
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).
DCR（Disease control rate） | 24months
  The percentage of cases with remission (PR + CR) and stable lesions (SD) after treatment was assessable.
DOR（Duration of response） | 24months
  DoR was defined as the time from the date of first documented response until the first date of documented progression or death in the absence of disease progression. The time of the initial response was defined as the latest of the dates contributing toward the first visit response of CR or PR. If a patient did not progress following a response, then their DoR was censored at the PFS censoring time.
OS (Overall survival time) | 24months
  The time of death from all causes for all patients from the date of randomization.
The Adverse Events | 24months
  AEs are any adverse medical events that occur in a subject or clinical subject and is not necessarily causally related to the treatment. Safety assessment in this study was conducted by the investigator in accordance with the definition of CTCAE 5.0.

IPD SHARING:
Plan to Share IPD: No